CLINICAL TRIAL: NCT01552993
Title: Registration and Treatment of Pain During Eye Examination of Prematurity
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: the chosen intervention was obviously ineffective
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HB2012-02
Record Dates: First submitted 2012-03-02; First posted 2012-03-13 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-04

CONDITIONS: Infant, Premature; Retinopathy
Keywords: prematurity; retinopathy; pain; acetaminophen
MeSH Terms: conditions — Premature Birth; Retinal Diseases; Pain | interventions — Acetaminophen; Sucrose

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- paracetamol (Experimental): Paracetamol mixture 20 mg/kg + pacifier and sucrose
  Interventions: Drug: paracetamol
- placebo (Placebo Comparator): pacifier and sucrose only
  Interventions: Drug: sucrose

INTERVENTIONS:
Drug: paracetamol — Paracetamol mixture 20 mg/kg + pacifier and glucose
  Arms: paracetamol
Drug: sucrose — pacifier and sucrose
  Arms: placebo

SUMMARY:
The aim of this study is to see if paracetamol has a pain-relieving effect during eye examination in premature infants.

DETAILED DESCRIPTION:
Retinopathy of prematurity (ROP) is a feared complication of premature birth. If discovered in time, the disease can be treated, and impaired vision or blindness can be reduced. Premature infants are therefore examined regularly after birth. However, the examination is painful and stressful for the infant. Painful experiences might lead to a pathological stress response later in life and should therefore be prevented.

This is a double blinded, controlled and randomized study where the infants are examined and assessed either with or without the use of paracetamol.

ELIGIBILITY:
Inclusion Criteria:

* Infants < 32 weeks of gestational age (< 31+6 weeks)

Exclusion Criteria:

* Infants with ongoing analgesic treatment

Ages: 31 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2012-03; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
pain | 5 minutes
  Premature Infant Pain Profile (PIPP): score range 0-21. Used independently by 2 experienced observers

CONTACTS AND LOCATIONS:
Overall Officials: Hakon Bergseng, PhD, Principal Investigator — St. Olavs University Hospital
Locations (1):
- St.Olavs University Hospital, Trondheim, Trøndelag, Norway